CLINICAL TRIAL: NCT07398625
Title: Management of Cesarean Section Scar Ectopic Pregnancy: Sohag University Experience
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Reem Kamel lotfy, Sohag, Sohag University
Other Study IDs: Soh-Med--25-4-11MS
Record Dates: First submitted 2025-05-11; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: CS Scar Pregnancy
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — observation of cs scar pregnancy cases &their management in Sohag University

SUMMARY:
management of CS scar ectopic pregnancy

ELIGIBILITY:
Inclusion Criteria:

1st trimester pregnancy (6-10) weeks Age: (18-40) years All types of scar ectopic pregnancy endophytic and exophytic types Viable and non-viable scar ectopic.

Exclusion Criteria:

Patients with serious systemic diseases will be excluded, such as; heart disease, thrombocytopenia, bronchial asthma and systemic lupus erythematosus because these conditions may affect treatment options and efficacy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1st trimester pregnancy (6-10) weeks Age: (18-40) years All types of scar ectopic pregnancy endophytic and exophytic types Viable and non-viable scar ectopic.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
irregular uterine bleeding and hematoma formation after surgical evacuation | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided